CLINICAL TRIAL: NCT01372826
Title: An Open-Label, Parallel-Group, Phase I Study to Compare the Pharmacokinetics of NKTR-118 Following a Single Oral Dose in Subjects With Renal Impairment and Subjects With Normal Renal Function
Brief Title: Assessing the Pharmacokinetics of NKTR-118 in Subjects With Renal Impairment Compared to That in Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3820C00009
Record Dates: First submitted 2011-05-25; First posted 2011-06-14 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Renal Impairment
Keywords: Phase 1; Pharmacokinetics; NKTR-118; renal impairment; parallel study; QTcF Interval; AUC(0-t); Cmax; tmax
MeSH Terms: conditions — Renal Insufficiency | interventions — naloxegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NKTR118 Group1 (Experimental): Normal Renal Function
  Interventions: Drug: NKTR118 Group1
- NKTR118 Group 2 (Experimental): Moderate Renal Function
  Interventions: Drug: NKTR118 Group 2
- NKTR118 Group 3 (Experimental): Severe Renal Impairment
  Interventions: Drug: NKTR118 Group3
- NKTR118 Group 4 (Experimental): End-Stage Renal Disease
  Interventions: Drug: NKTR118

INTERVENTIONS:
Drug: NKTR118 Group1 — Oral dose, 25 mg
  Arms: NKTR118 Group1
Drug: NKTR118 Group 2 — Oral dose, 25 mg
  Arms: NKTR118 Group 2
Drug: NKTR118 Group3 — Oral dose, 25 mg
  Arms: NKTR118 Group 3
Drug: NKTR118 — Oral dose, 25 mg
  Arms: NKTR118 Group 4

SUMMARY:
This study will be assessing the pharmacokinetics of NKTR-118 in subjects with renal impairment compared to that in subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written and dated informed consent prior to any study specific procedures.
* Male or female volunteers aged 18 to 80 years (inclusive) having normal renal function, or suffering from moderate or severe renal impairment or ESRD.

Male subjects who are sexually active must be willing to use a barrier method of contraception (condom). Women must be of non-childbearing potential or, if of childbearing potential, must have a negative pregnancy test (at screening and at each admission) and be using a highly effective form of birth control for 3 months before enrollment and be willing to use a highly effective form of birth control during the study and until 3 months after their last dose of IP.

* Have a BMI between 18 and 40 kg/m2 (inclusive) and weigh at least 50 kg.
* Subjects must be able to understand and to comply with study procedures, restrictions and requirements.

Exclusion Criteria:

* History of any clinically significant medical history which, in the opinion of the Investigator and Sponsor, may either put the subject at risk because of participation in the study, or influence the results, or the subject's ability to participate in the study.
* History or presence of gastrointestinal hepatic or other condition known to interfere with disposition of the study drug (except for renal function impairment).
* Subjects who have a functioning kidney transplant.
* Acute illness, surgical procedures or trauma from within 2 weeks before enrollment until first administration of study drug
* Known or suspected history of drug abuse as judged by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of a single dose of NKTR-118 25 mg by assessment of area under the curve over the time (AUC) | PK blood samples will be collected in treatment periods 1 and 2 at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 h post-dose.
  Groups 1 (normal), 2 (moderate), 3 (severe), and for Group 4 (End-stage renal disease requiring hemodialysis)
To assess the pharmacokinetics of a single dose of NKTR-118 25 mg by assessment of maximum concentration (Cmax) | PK blood samples will be collected in treatment periods 1 and 2 at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 and 72 h post-dose.
  Groups 1 (normal), 2 (moderate), 3 (severe), and for Group 4 (End-stage renal disease requiring hemodialysis)

SECONDARY OUTCOMES:
To assess the safety and tolerability of NKTR-118 in subjects with renal impairment and normal renal function by assessing Adverse events. | Duration Day -1 to follow-up at either visit 3 or 6 dependant on treatment
To assess the safety and tolerability of NKTR-118 in subjects with renal impairment and normal renal function by assessing vital signs | Duration Day -1 to follow-up at either visit 3 or 6 dependant on treatment
To assess the safety and tolerability of NKTR-118 in subjects with renal impairment and normal renal function by assessing safety blood samples | Duration Day -1 to follow-up at either visit 3 or 6 dependant on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center US
Locations (3):
- United States (3):
  - Research Site, Anaheim, California
  - Research Site, Orlando, Florida
  - Research Site, Overland Park, Kansas

REFERENCES:
- [Derived] Bui K, She F, Sostek M. The effects of renal impairment on the pharmacokinetics, safety, and tolerability of naloxegol. J Clin Pharmacol. 2014 Dec;54(12):1375-82. doi: 10.1002/jcph.349. Epub 2014 Jul 1. PMID 24946021
- See also: D3820C00009 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1391&filename=D3820C00009_Clinical_Study_Report_Synopsis.pdf